CLINICAL TRIAL: NCT03248687
Title: Home Management Versus Primary Care Physician Follow up in Children With Distal Radius Fractures: A Randomized Control Trial
Brief Title: Distal Radius Buckle Fracture Follow up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Physician Services Incorporated (Unknown)
Responsible Party: Principal Investigator, Kathy Boutis, Staff Physician and Sr. Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000053044
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized to one of two follow up arms
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know if the patient was followed at home or by a primary care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home follow up (Experimental): Patients with a distal radius buckle fracture treated in a removable splint will be provided with discharge instructions and anticipatory guidance without any scheduled physician follow up.
  Interventions: Other: Follow up
- Primary Care Physician Follow up (Active Comparator): Patients with a distal radius buckle fracture treated in a removable splint will be provided with discharge instructions and anticipatory guidance with scheduled primary care physician follow up at 1-2 weeks post visit to the emergency department.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — The intervention will be method of follow up.

SUMMARY:
The investigators will be enrolling children with distal radius buckle fractures, treating them with a removable splint and randomizing them to follow up as needed vs required follow up with a primary care physician 1-2 weeks after the ED visit.

DETAILED DESCRIPTION:
Buckle fractures of the distal forearm that include the radius are the most common fracture in childhood, and the risk of this fracture occurring is about 1 in every 25 children.Despite the high frequency of this fracture, it is a very stable injury and thus can be safely treated with a removable wrist splint while the fracture heals. Furthermore, authors have concluded that since orthopedic intervention is exceedingly rare, this type of fracture may safely be followed by a primary care physician (PCP) or managed at home.

In Canada, about 50% of these injuries are routinely discharged from the ED for follow up with the PCP, instead of an orthopedic clinic. The investigators' work examined the management outcomes of 180 children with a distal radius buckle fractures who were treated in an ED with a removable splint, given anticipatory guidance, and advised to follow up in two weeks with their PCP. We demonstrated that PCP follow up was safe and effective, with about 90% of patients completing their care at the PCP without additional visits to an ED or orthopedic surgeon. All patients recovered as expected without complications. However, about 50% of these patients did not receive additional anticipatory guidance from their PCPs on duration of splint use or expected timing of return to usual activities at the PCP visit. Nevertheless, patients with and without this additional anticipatory guidance reported a similar duration of splint use and timing for return to usual activities, largely based on what was recommended at the ED visit. Since these injuries are inherently stable, carry an excellent prognosis, and are treated with a splint that can be removed at home in accordance with anticipatory guidance provided in the ED, it calls into question the need for any routine physician follow up of these common minor fractures.

If home management of distal radius buckle fracture after ED discharge demonstrated safety and effectiveness in a methodologically robust study, it would have clear advantages for patients and families, physicians, and the health care system. The frustrations of lengthy clinic visits and transport difficulties would be avoided. Parents would miss less time away from work or other priorities, and the patients themselves would not miss school. In medically under-serviced communities in particular, patients would avoid long travel distances to see a physician for this minor injury where physician intervention after the ED visit is rarely required. Furthermore, it will obviate the need to shift the care of these common minor fractures from the orthopedic surgeon to the PCP, relieving some pressure on health care practitioners and increase availability for other patients more in need of physician services. Importantly, the potential for reduced use of superfluous health care services for this common injury is also likely to result in health care cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy children aged 5 to 17 years who present to the study ED within three days of a wrist injury that is diagnosed in the ED as a distal radius buckle fracture will be eligible for enrolment. Furthermore, approximately 15% of children with this fracture have an associated ulnar buckle or ulnar styloid fracture. In previous similar research, children with these associated ulnar fractures were included in the study population. Thus, distal radius buckle fractures with or without an associated buckle/styloid fracture of the distal ulna will be eligible for participation.

Exclusion Criteria:

1. Children at risk for pathologic fractures such as those with congenital or acquired bony disease (Appendix I).
2. Congenital anomalies of the extremities which may complicate clinical or radiographic assessment.
3. Multisystem trauma and multiple fractures of the same limb since these patients would require additional management and follow-up beyond that of an isolated buckle fracture.
4. Patients cognitively and developmentally delayed such that they are unable to communicate pain or have limited performance in activities of daily living at baseline.
5. Past history of ipsilateral distal radius/ulna fracture within 3 months of enrollment.
6. Patients who do not have phone or electronic mail access. This will preclude follow up of these patients.
7. Patients in whom the English language is so limited that consent and/or follow up is not possible.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Activity Scales for Kids - Performance Version, which is a validated activity scale that measures the ability of a child's physical function | Three weeks post injury
  The Activity Scales for Kids is a validated activity scale that measures a child's physical function

SECONDARY OUTCOMES:
Proportion of children with splint use "almost all of the time" > 3 weeks duration | 12 weeks
  The investigators will ask parents at three weeks if they use the splint, "almost never," "sometimes," "frequently," or "almost all of the time."
Proportion of children who received unscheduled visits to a physician for the index wrist injury, obtained by parental report and Canadian Institute of Health Information data | 12 weeks
  At 12 weeks, the investigators will determine which children visited a physician for the index wrist injury as per parental report and/or data available from CIHI
Proportion of parents who rated the satisfaction with their care as "very satisfied/satisfied." | 4 weeks
  The investigators will ask parents to rate the satisfaction with their care at 4 weeks on the following scale: "unsatisfied," somewhat satisfied," and "very satisfied."
Health Economic Evaluation - dollar values will be obtained for patient and health care costs and compared between the groups. | 12 weeks
  The investigators will determine costs of patient and health care events using available sources for this information.

CONTACTS AND LOCATIONS:
Locations (1):
- Kathy Boutis, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colaco K, Willan A, Stimec J, Barra L, Davis A, Howard A, Boutis K. Home Management Versus Primary Care Physician Follow-up of Patients With Distal Radius Buckle Fractures: A Randomized Controlled Trial. Ann Emerg Med. 2021 Feb;77(2):163-173. doi: 10.1016/j.annemergmed.2020.07.039. Epub 2020 Oct 21. PMID 33500115